CLINICAL TRIAL: NCT01466465
Title: Vitamin D and Grass Pollen Specific Immunotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Margitta Worm, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ProGIT; 2010-021775-80 (EudraCT Number)
Record Dates: First submitted 2011-11-01; First posted 2011-11-08 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Vitamin D; SIT; Grass pollen; allergic rhinoconjunctivitis
MeSH Terms: interventions — Cholecalciferol; Vitamin D; Carrier State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vigantol (Experimental)
  Interventions: Drug: Cholecalciferol
- neutral oil (vigantol carrier) (Placebo Comparator)
  Interventions: Other: middle-chain fatty acids (carrier)

INTERVENTIONS:
Drug: Cholecalciferol — given orally, once daily, before grass pollen season
  Other Names: Vitamin D
  Arms: Vigantol
Other: middle-chain fatty acids (carrier) — given orally, once daily, before grass pollen season
  Other Names: neutral oil
  Arms: neutral oil (vigantol carrier)

SUMMARY:
Allergen-specific immunotherapy is the only causal therapy of Immunoglobulin E-induced allergies like allergic rhinoconjunctivitis. Despite progress during the last decades it is limited by a long treatment time and high non-responder frequency. Based on experimental and epidemiological evidences we hypothesize that vitamin D can act as an effective immunomodulatory adjuvant to overcome these limitations.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* relative Vitamin D deficiency
* clinical relevant grass pollen allergy
* positive intradermal test with grass pollen
* forced expiratory volume at one second (FEV1) > 70%

Exclusion Criteria:

* current specific immunotherapy
* instable allergic asthma
* pregnancy and lactation
* treatment with immunomodulators or immunosuppressive drugs
* sarcoidosis, chronic diseases, malignancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
wheal diameter in the intradermal test after SIT in the comparison between vitamin D and placebo | three years

CONTACTS AND LOCATIONS:
Overall Officials: Worm Margitta, MD, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Allergy-Centre-Charité, CCM, Berlin, Germany